CLINICAL TRIAL: NCT03143530
Title: The Effect of Pectoralis Block on Analgesia After Simple Mastectomy
Brief Title: Effect of Pectoralis Block on Analgesia After Simple Mastectomy
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Extensive protocol revisions initiated.
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: Duke University (Other)
Responsible Party: Principal Investigator, Uma Shastri, Assistant Professor of Anesthesiology, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 160419
Record Dates: First submitted 2017-03-20; First posted 2017-05-08 (Actual); Last update posted 2018-08-14 (Actual); Status verified 2018-08

CONDITIONS: Mastectomy; Nerve Block; Analgesia, Postoperative
Keywords: Ropivacaine
MeSH Terms: conditions — Agnosia | interventions — Saline Solution; Ropivacaine

STUDY DESIGN:
Intervention Model Description: Participants will be assigned to one of two of the following groups for the duration of the study.
  1. General anesthesia + pectoralis block with Ropivacaine 30ml of 0.25% (75mg)
  2. General anesthesia + sham block with 30ml of normal saline
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants, care providers, investigators, and observers who record central measurements will be blinded to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pectoralis Block with Ropivacaine (Active Comparator): General anesthesia + pectoralis block with ropivacaine injection 30ml of 0.25% (75mg)
  Interventions: Procedure: Pectoralis block; Drug: Ropivacaine Injection
- Pectoralis Block with normal saline (Placebo Comparator): General anesthesia + Pectoralis block with 30ml of normal saline injection
  Interventions: Procedure: Pectoralis block; Drug: Normal saline injection

INTERVENTIONS:
Procedure: Pectoralis block — Pectoralis block involving injection near the coracoid process in the fascial planes between both the pectoralis major and minor muscles (pecs I), and the fascial plane between the pectoralis minor and serratus anterior muscles (pecs II).
Drug: Normal saline injection — Pectoralis block involving injection of normal saline 30ml near the coracoid process in the fascial planes between both the pectoralis major and minor muscles (pecs I), and the fascial plane between the pectoralis minor and serratus anterior
  Arms: Pectoralis Block with normal saline
Drug: Ropivacaine Injection — Pectoralis block involving injection of ropivacaine injection 30ml of 0,25% (75 mg) near the coracoid process in the fascial planes between both the pectoralis major and minor muscles (pecs I), and the fascial plane between the pectoralis minor and serratus anterior
  Arms: Pectoralis Block with Ropivacaine

SUMMARY:
The pectoralis block, including pecs I and II block, is a novel technique first described in 2011 as an alternative to paravertebral blockade for analgesia following breast surgery. The research goal is to determine the efficacy of the pectoralis block compared to placebo in improving quality of recovery following mastectomy.

DETAILED DESCRIPTION:
The pectoralis block, including pecs I and II block, is a novel technique first described in 2011 as an alternative to paravertebral blockade for analgesia following breast surgery. The concept involves injecting local anesthetic near the coracoid process in the fascial planes between both the pectoralis major and minor muscles (pecs I), and the fascial plane between the pectoralis minor and serratus anterior muscles (pecs II). This is a prospective, double-blinded, randomized controlled trial in subjects undergoing mastectomy under general anesthesia. The research goal is to determine the efficacy of the pectoralis block compared to placebo in improving quality of recovery following mastectomy.

ELIGIBILITY:
Inclusion Criteria:

* ASA 1, 2, and 3 patients (According to ASA classification of comorbid conditions and general health)
* Patients undergoing simple mastectomy

Exclusion Criteria:

* -Patient Refusal
* Allergy to local anesthetics
* Inability to communicate in English
* Use of 8 mg morphine equivalents or greater currently and for a period of longer then 2 weeks prior to surgery
* Existing nerve injuries or sensory deficits
* Conversion to anesthesia via an endotracheal tube

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-12 (Estimated); Primary Completion 2019-03-01 (Estimated); Study Completion 2019-04-01 (Estimated)

PRIMARY OUTCOMES:
Quality of Recovery-27 score at baseline | Baseline
  Quality of Recovery-27 score, a validated tool to assess quality of postoperative recovery at baseline
Quality of Recovery-27 score at post operative day 1 | Post operative day 1
  Quality of Recovery-27 score, a validated tool to assess quality of postoperative recovery, at baseline and post operative day 1
Quality of Recovery-27 scores at post operative day 7 | Post operative day 7
  Quality of Recovery-27 score, a validated tool to assess quality of postoperative recovery, at baseline and post operative day 7
Quality of Recovery-27 scores at post operative day 30 | Post operative day 30
  Quality of Recovery-27 score, a validated tool to assess quality of postoperative recovery, at baseline and post operative day 30
Quality of Recovery-27 scores at post operative day 90 | Post operative day 90
  Quality of Recovery-27 score, a validated tool to assess quality of postoperative recovery, at baseline and post operative day 90

SECONDARY OUTCOMES:
Comparison of Numerical Rating Scale-11 (NRS-11) at rest | 90 days
  Comparison of patient reported pain assessment while at rest using the NRS-11 Scale at arrival in PACU, 15 minutes, 30 minutes, 1 hour and 2 hours after arrival in PACU, and postoperative days 1, 7, 30, and 90. The NRS-11 is a 11 point scale when 0 is no pain and 10 is severe pain.
Comparison of Numerical Rating Scale-11 (NRS-11) with movement | 90 days
  Comparison of patient reported pain assessment while with movement using the NRS-11 Scale at arrival in PACU, 15 minutes, 30 minutes, 1 hour and 2 hours after arrival in PACU, and postoperative days 1, 7, 30, and 90. The NRS-11 is a 11 point scale when 0 is no pain and 10 is severe pain.
Duration of postoperative analgesia | Up to 24 hours
  Duration of postoperative analgesia as measured by time in minutes to first intravenous or oral opioid postoperatively.

CONTACTS AND LOCATIONS:
Overall Officials: Uma Shastri, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No